CLINICAL TRIAL: NCT00389662
Title: The Effect of Wearing the 'Nike Free'Shoe on Isokinetic Muscle Strength of Foot and Ankle and on Proprioception.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Ghent (Other)
Collaborators: Nike (Industry)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2006/345
Record Dates: First submitted 2006-10-18; First posted 2006-10-19 (Estimated); Last update posted 2007-12-28 (Estimated); Status verified 2007-12

CONDITIONS: Healthy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: Wearing the "Nike Free" shoe

SUMMARY:
To evaluate the effect of wearing the 'Nike Free'Shoe on isokinetic muscle strength of foot and ankle and on proprioception the following protocol will be used.

The test population consists out of students of the physical education department. They will at random be divided in three groups. One group will wear the shoe only for daily activities, the second group will wear the shoes for the warming up part of the sport classes and the control group will not wear the shoe at all. There will be two moments for evaluation: one at the beginning of the study and one after four months, during which the shoe will be used. The isokinetic strength will be measured with an isokinetic device (Biodex) and the proprioception will be evaluated with a force platform (Neurocom Balance Master).

ELIGIBILITY:
Inclusion Criteria:

* being a physical education student of the second or third year
* having read and signed the informed consent
* being new to the Nike Free Shoe

Exclusion Criteria:

* neurological or systemic diseases
* overuse injuries or orthopaedic surgery to the lower limbs during the previous six months
* familiar to or used to wear the Nike Free Shoe

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 45 (Estimated)
Dates: Start 2006-11; Study Completion 2007-04 (Actual)

PRIMARY OUTCOMES:
Isokinetic strength of foot and ankle muscles and on proprioception | 4 months after starting the data registration

CONTACTS AND LOCATIONS:
Overall Officials: Philip Roosen, Physiotherapist, Principal Investigator — University Ghent
Locations (1):
- University Ghent, Ghent, Belgium

REFERENCES:
- See also: Website University Ghent — http://www.ugent.be